CLINICAL TRIAL: NCT01856426
Title: Double-Blind, Randomized, Placebo-controlled, Multi-center Trial to Determine the Safety and Antiviral Effect of Single Doses of EDP239 in Hepatitis C Virus (HCV) Infected Subjects
Brief Title: Proof of Concept Study for Safety and Efficacy of EDP239 in Hepatitis C Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEDP239X2201
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C
Keywords: Hepatitis C infected subjects
MeSH Terms: conditions — Hepatitis C | interventions — EDP-239

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1- EDP239 (Experimental): EDP239 given once a day.
  Interventions: Drug: EDP239
- Placebo (Placebo Comparator): 1 treatment arm will be placebo, dose given once a day.
  Interventions: Drug: Placebo
- 2- EDP239 (Experimental): EDP239 given once a day.
  Interventions: Drug: EDP239
- 3-EDP239 (Experimental): EDP239 given once a day.
  Interventions: Drug: EDP239
- 4-EDP239 (Experimental): EDP239 given once a day.
  Interventions: Drug: EDP239

INTERVENTIONS:
Drug: EDP239
  Arms: 1- EDP239; 2- EDP239; 3-EDP239; 4-EDP239
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is, to assess whether EDP239 can reduce the HCV viral load in HCV gentotype-1 in chronically infected subjects and to further evaluate the safety profile of EDP239.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have chronic genotype-1 hepatitis C virus infection and plasma HCV-RNA ≥ 105 IU/mL at the time of screening.
* Subjects must have chronic HCV infection as determined by any of the following:
* be anti-HCV (+) for at least 6 months per subject history or medical records
* an anti-HCV test, viral load, or genotype > 6 months ago
* In the setting of a recent positive anti-HCV test (< 6 months), liver biopsy demonstrating chronicity
* Subjects must have IL-28b genotype "CC"
* Subjects must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 36 kg/m2. BMI = Body weight (kg) / [Height (m)]2

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days (for small molecules) whichever is longer; or longer if required by local regulations.
* Previous treatment, including the use of any investigational agents, for the treatment of HCV infection.
* Women of child bearing potential.
* Subjects with IL-28b genotype "CT or TT".
* ALT γ-GT, and AST must be below 5 x the upper limit of normal (ULN).
* Serum bilirubin must not exceed ULN.
* The PT (INR) must be within normal limits.
* If necessary, laboratory testing may be repeated on one occasion (as soon as possible) prior to randomization, to rule out any laboratory error.
* Use of drugs that inhibit or induce CYP3A4.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline Hepatitis C viral load at Day 1 | baseline, day 1
  Blood will be collected for Hepatitis C viral load at Day 1.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety | 14 days
  Laboratory and clinical evaluations will be used as safety events
Change from baseline in HCV RNA log | baseline, Day 1
  A viral load drop in excess of 2.5 will be considered a success.
Total concentration in plasma of EDP239 in HCV Gentoype 1 infected subjects | baseline, day 1
  The concentration in plasma parameters of EDP239 will be determined using the actual recorded sampling times and non-compartmental method.

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Study Director — Enanta Pharmaceuticals, Inc
Locations (5):
- United States (3):
  - Investigative Site, Miami, Florida
  - Investigative Site, San Antonio, Texas
  - Investigative Site, Murray, Utah
- Germany (2):
  - Investigative Site, Frankfurt
  - Investigative Site, Hamburg

REFERENCES:
- [Derived] Owens CM, Brasher BB, Polemeropoulos A, Rhodin MH, McAllister N, Wong KA, Jones CT, Jiang L, Lin K, Or YS. Preclinical and Clinical Resistance Profile of EDP-239, a Novel Hepatitis C Virus NS5A Inhibitor. Antimicrob Agents Chemother. 2016 Sep 23;60(10):6216-26. doi: 10.1128/AAC.00815-16. Print 2016 Oct. PMID 27503644
- [Derived] Owens CM, Brasher BB, Polemeropoulos A, Rhodin MH, McAllister N, Peng X, Wang C, Ying L, Cao H, Lawitz E, Poordad F, Rondon J, Box TD, Zeuzem S, Buggisch P, Lin K, Qiu YL, Jiang L, Colvin R, Or YS. Preclinical Profile and Clinical Efficacy of a Novel Hepatitis C Virus NS5A Inhibitor, EDP-239. Antimicrob Agents Chemother. 2016 Sep 23;60(10):6207-15. doi: 10.1128/AAC.00808-16. Print 2016 Oct. PMID 27503640